CLINICAL TRIAL: NCT01534949
Title: A Phase 1, Multicenter, Open-Label, Single-Arm Study to Evaluate the Initial Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of CT-P10 Given in Combination With Dexamethasone, Cytosine Arabinoside, and Cisplatin (DHAP) in Patients With Diffuse Large B-Cell Lymphoma as Second-Line Chemotherapy
Brief Title: Provide Initial Evidence of Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy to Support the Pivotal CT-P10 Therapeutic Equivalence Trial
Acronym: Triad-DLBCL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-P10 1.2
Record Dates: First submitted 2012-02-08; First posted 2012-02-17 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL, Biosimilar
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT-P10 (Experimental): rituximab
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — 375 mg/m2 by intravenous [IV] infusion

SUMMARY:
This study is designed to provide initial evidence of safety, pharmacokinetics, pharmacodynamics, and efficacy to support the pivotal CT-P10 therapeutic equivalence trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically proven DLBCL, which may represent de novo DLBCL or DLBCL arising from transformed follicular lymphoma or chronic lymphocytic leukemia.
2. Patient has relapsed or refractory CD20-positive disease following previous first-line systemic chemotherapy. Patients who have failed to achieve complete remission with previous chemotherapy are defined as refractory, and those who relapsed after an initial complete remission are classified as having relapsed. A biopsy must be performed to confirm diagnosis of relapsed disease. Tumor tissue within 6 months of Day 1 of Cycle 1 of study treatment will be used for the central review.
3. Patient has at least 1 measurable tumor mass (greater than 1.5 cm in the longest dimension, or 1.1 to 1.5 cm in the longest dimension, and greater than 1.0 cm in the shortest axis) that has not previously been irradiated or has grown since previous irradiation

Exclusion Criteria:

1. Patient has allergies or hypersensitivity to murine, chimeric, human, or humanized proteins.
2. Patient has had prior allogeneic or ASCT.
3. Patient has received any other anticancer therapy within 28 days before Day 1 of Cycle 1 of study treatment and more than 1 prior line of chemotherapy, with the exception of having received the last dose of rituximab within 6 months before Day 1 of Cycle 1 of study treatment if they have undergone prior treatment with rituximab.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
safety | after 6 weeks of treatment begin
  Adverse events, including SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Wonseog Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea